CLINICAL TRIAL: NCT06836739
Title: At-Home Feasibility Trial of Genital Nerve Stimulation to Modulate Neurogenic Bowel Dysfunction in Individuals Living With Spinal Cord Injury
Brief Title: At-Home Genital Nerve Stimulation for SCI Bowel
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: MetroHealth Medical Center (Other)
Collaborators: Congressionally Directed Medical Research Programs (U.S. Federal Agency)
Responsible Party: Principal Investigator, Kimberly Anderson, PhD, Professor, MetroHealth Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY00000717; W81XWH2210778 - SC210121 (Other Grant/Funding Number: Department of Defense CDMRP SCIRP); W81XWH2210781 - SC210121P1 (Other Grant/Funding Number: Department of Defense CDMRP SCIRP)
Record Dates: First submitted 2025-01-31; First posted 2025-02-20 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Spinal Cord Injury
Keywords: fecal incontinence; neurogenic bowel; tetraplegia; paraplegia; paralysis; electrical stimulation; neuromodulation; bowel; feasibility; anorectal manometry
MeSH Terms: conditions — Spinal Cord Injuries; Fecal Incontinence; Neurogenic Bowel; Quadriplegia; Paraplegia; Paralysis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Target genital nerve stimulation (Experimental): Stimulation waveforms consist of biphasic, charge-balanced square pulses with a pulse width of 0.2 ms and delivered at 20 Hz. Stimuli will be applied over a range of amplitudes to determine the threshold of stimulation for producing reflex contraction of the anal sphincter (the pudendo-anal reflex). Subsequent stimulation will be applied at threshold for the first week, at 1.5 threshold for the second week, and at twice threshold (or max tolerance) for the third and fourth weeks. The typical stimulation range is 20-40 milliamps (mA) and has been shown to be well tolerated by individuals with sensation. Stimulation will be applied continuously for 6-8 hours daily for four weeks.
  Interventions: Device: Genital nerve stimulation
- Sham genital nerve stimulation (Sham Comparator): Sham stimulation will be applied in the same manner as target stimulation, except that the stimulation frequency will be 1 Hz and the stimulation amplitude will be set to a limit that is at the threshold of perception if individuals have sensation, or 10 mA if they do not have sensation. Stimulation will be applied continuously for 6-8 hours daily for four weeks.
  Interventions: Device: Genital nerve stimulation

INTERVENTIONS:
Device: Genital nerve stimulation — Genital nerve stimulation (GNS) will be administered via non-invasive surface skin electrodes. In men, two surface electrodes (1 cm diameter) will be placed on the dorsum of the penile shaft 2 cm apart. In women, one surface electrode will be placed near the clitoris and a second surface electrode will be placed on the labia majora or inner thigh. The electrodes will be connected to an electrical stimulator device.

SUMMARY:
The purpose of this study is to test whether electrical stimulation of the skin in the pelvic area (near the genitals) can reduce the reflexes that cause bowel accidents in people with spinal cord injuries. Current bowel treatments either involve diet and medications or surgery. This study will evaluate whether electrical stimulation can be an alternate option for bowel management.

Researchers will:

* Use an FDA approved Transcutaneous Electrical Nerve Stimulation (TENS) device off-label
* Compare a target stimulation level to a placebo stimulation level

Participants will:

* Use electrical stimulation on the skin in the pelvic area for 6-8 hours each day for 4 weeks at home
* Visit the research center 3 times to participate in exams and answer questions
* Keep a daily diary of their bowel symptoms and stimulation times

DETAILED DESCRIPTION:
The objective of this proposal is to determine how genital nerve stimulation (GNS) acutely modulates neurogenic bowel dysfunction (NBD) in individuals with different severities of spinal cord injury (SCI) and to determine the key study design and methodology parameters of daily at-home administration of GNS. This study will determine the feasibility of daily application of GNS as an intervention for NBD. Key feasibility measures related to dosage and adherence will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

1. Traumatic SCI.
2. Minimum of 6 months' post-injury.
3. Aged 18 years and older.
4. Neurological level of injury T12 or higher and AIS grade A-D, as defined by the ISNCSCI.
5. Score of 14 or higher on the ISCI BF BDS v2.1.
6. Response to genital nerve stimulation able to be elicited upon screening.
7. Able to understand and provide informed consent.

Exclusion Criteria:

1. Currently enrolled in another functional electrical stimulation (FES) research trial.
2. Females who are pregnant or planning to become pregnant in the duration of the trial (identified by self-report).
3. Presence of a cardiac pacemaker, implanted defibrillator, or other implanted functional electrical stimulation device if, upon clinical evaluation, it may have an interaction with GNS.
4. In the judgment of the PI and Co-Investigators, presence of medical complications that may interfere with the execution of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2025-03-01 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
The primary endpoint will be the feasibility of daily application of GNS as an intervention for NBD. | From baseline to the end of 6 weeks
  The 1st feasibility measure bench mark will be the proportion of enrolled who complete the full stimulation protocol.
The primary endpoint will be the feasibility of daily application of GNS as an intervention for NBD. | From baseline to the end of 6 weeks
  The 2nd feasibility measure bench mark will be the number of occurrences of unblinding.
The primary endpoint will be the feasibility of daily application of GNS as an intervention for NBD. | From baseline to the end of 6 weeks
  The 3rd feasibility measure bench mark will be the retention rate.

SECONDARY OUTCOMES:
Anorectal Manometry (ARM) | From baseline to the end of 6 weeks
  The main secondary endpoint will be anorectal reflex activity as measured by ARM. ARM is the gold standard clinical tool for investigating anorectal function. It is widely available and very well established. Recent efforts have been made to standardize ARM testing protocols so that results can be categorized. The London Classification protocol will be used in ARM testing in this experiment.
Clinical exam | From baseline to the end of 6 weeks
  This is conducted by a clinician and involves a gastrointestinal system clinical exam of bowel dysfunction.
Bowel diary | From baseline to the end of 6 weeks.
  A bowel diary is a means for participants to record daily bowel activities. It will be time-stamped. Parameters that are targeted to be recorded include stool type (using the Bristol Stool Scale), amount, planned emptying episodes (including time), incontinence episodes, sense of urgency, straining, medications, and complications such as nausea or hemorrhoids. These data will characterize each participant's bowel management routine, daily habits, and gastrointestinal (GI) symptoms.
Stimulation diary | From baseline to the end of 6 weeks.
  A record of hours of daily stimulation use will also be captured in a stimulation diary.
International SCI (ISCI) Bowel Function (BF) Basic Dataset (BDS) version 2.1 | From baseline to the end of 6 weeks.
  The ISCI BF BDS v2.1 incorporates the Neurogenic Bowel Dysfunction Score as well as information about GI or anal sphincter dysfunction unrelated to SCI, surgical procedures on the GI tract, defecation methods and bowel care procedures, the need to wear external continence products, and presence of abdominal pain or discomfort. The NBDS was developed specifically for SCI and measures the degree of neurogenic bowel dysfunction symptomology and the impact on quality of life (QoL). There are 10 items, and they are symptom-based and weighted by the impact on QoL. The score ranges from 0-45 with a higher score meaning a worse outcome.
SCI-QoL Bowel Management Difficulties (SCI-QoL BMD) | From baseline to the end of 6 weeks.
  The SCI-QoL BMD measures difficulties people living with SCI have with bowel management, including feelings of distress associated with bowel problems they experience in daily life. The items focus on issues related to fecal incontinence and the psychosocial consequences of fecal incontinence, which is different that the ISCI BF BDS v2.1 and why it was selected as an additional secondary outcome measure. The full scale is composed of 26 items, but a computer assisted technology version and 9-item short form version have also been created. The short form version will be used in this trial and is available for download from Assessment Center. Each item has a response option based on a 5-point Likert scale ranging from 1 'never/not at all' to 5 always/very much'. Raw scores range from 9-45 with higher scores representing greater difficulty managing bowel problems.
SCI Common Data Elements (CDEs) | At baseline.
  SCI CDEs to be collected include 1) Medical History for body system categories including start date, end date, and ongoing status, 2) History of Injury (injury time frame, injury etiology), 3) Demographics (gender, birth date, race, ethnicity, marital status, number of members in household, area of residence, number of years of education, primary occupation), and 4) International Standards for Neurological Classification of SCI for injury classification (upper extremity motor score, lower extremity motor score, total motor score, light touch sensory score, pinprick sensory score, deep anal pressure, voluntary anal contraction, zone of partial preservation, and impairment grade data)

OTHER OUTCOMES:
Treatment questionnaire | At the end of 6 weeks.
  It is important to be able to collect participant feedback on the ease or difficulty of using the TENS unit and applying GNS at home. This is important feasibility information that should be collected, and we will generate a form to enable more standardized collection of this data from each participant. This will include prompts such as any difficulty placing electrodes, any difficulty keeping electrodes in place, any need for further training on the device once home, any device malfunctions, any need for replacement components or electrodes, etc.
Study exit questionnaire | At the end of 6 weeks.
  A study exit questionnaire will be used to determine whether participants remained blinded throughout the study and any perspectives on their experience while in the study.

CONTACTS AND LOCATIONS:
Overall Officials: Kim Anderson, PhD, Principal Investigator — MetroHealth System, Ohio
Locations (1):
- MetroHealth Center for Rehabilitation Research, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: Yes
A deidentified dataset will be transferred to the Inter-University Consortium for Political and Social Research (ICPSR) for data sharing and long-term preservation.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Within 12 months of the end of study.
Access Criteria: Based on ICPSR guidelines.

DOCUMENTS (1):
  • Informed Consent Form (2025-08-08): https://cdn.clinicaltrials.gov/large-docs/39/NCT06836739/ICF_002.pdf